CLINICAL TRIAL: NCT04071535
Title: Application of Skin Biopsy in the Early Diagnosis of Small Fiber Neuropathy in Chinese Patients With Diabetes
Brief Title: Skin Biopsy in the Diagnosis of Small Fiber Neuropathy in Chinese Patients With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: SFNChinaDM
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Small Fiber Neuropathy; Diabetic Neuropathies; Diabetes Mellitus
Keywords: Small fiber neuropathy; Diabetic neuropathies; Skin biopsy
MeSH Terms: conditions — Small Fiber Neuropathy; Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Skin sample, blood serum (approximately 3ml), and whole blood (approximately 6ml).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sudoscan、nerve conduction tests — To evaluate sudomotor nerve and macrofibropathy.

SUMMARY:
To detect small fiber neuropathy in patients with possible or established diabetic peripheral neuropathy (DPN) by skin biopsy and explore clinical characteristics and pathological features in Chinese patients with diabetes.

DETAILED DESCRIPTION:
Small fiber neuropathy (SFN) is a subtype of diabetic neuropathy, patients with SFN often manifest as paresthesia of warmth, cold, pinprick and so on, especially affect ed length-dependent area. Skin biopsy is an effective method to diagnose SFN with high diagnostic accuracy. The procedure is simple and minimally, and the wound usually heals within a few days. However, skin biopsy is not widely used in diagnose of SFN in Chinese patients with diabetes. This study is aimed to establish a normal reference range of intraepidermal nerve fiber density (IENFD) in the Chinese population, and to detect SFN in Chinese patients with diabetes by skin biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18 and ≦75 years old
* A history of diabetes
* Symptoms of small fiber neuropathy such as pain, paresthesia, acanthesthesia after diagnosed with diabetes

Exclusion Criteria:

* Acute skin infection or injury
* Coagulation disorders
* History of malignant tumor
* Usage of neurotoxic drugs
* Alcohol abuse
* Vascular diseases, e.g. LEASO and stroke
* Infectious diseases, e.g. hepatitis B, HIV, and syphilis
* Metabolic disorders, e.g. hypothyroidism, hyperlipidemia, and amyloid lesions
* Connective tissue diseases
* Nutritional disorders, e.g.vitamin B6 deficiency, and vitamin B12 deficiency
* Other causes of peripheral neuropathy, e.g. lumbar disc herniation, Guillain-Barre Syndrome, and polyradiculopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese patients complaining symptoms of neuropathies after diagnosed diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of small fiber neuropathy in Chinese patients with diabetes by calculating intraepidermal nerve fiber density (IENFD) via skin biopsy | December, 2019
  Calculating intraepidermal nerve fiber density (IENFD) is considered as as gold criteria of diagnosis of small fiber neuropathy.

SECONDARY OUTCOMES:
Evaluation of diagnostic sensitivity and specificity of sudoscan in Chinese diabetic patients with small fiber neuropathy compared with intraepidermal nerve fiber density (IENFD) | December, 2019
  Sudoscan is used to as an autonomic nerve assessment tool with objective and stable operations, which measures the function of sweat glands by stimulating a low voltage current ( < 4 volts) and detects the electrochemical reaction between the electrodes and chloride ions in both hands and feet. Results are presented as electrochemical skin conductance in hands (HESC) and feet (FESC), asymmetry ratio value in hands (HASYM) and feet (FASYM). We use intraepidermal nerve fiber density (IENFD) measured by skin biopsy as the gold standard, sudoscan is used to evaluate its diagnostic efficiency including sensitivity and specificity of small fiber neuropathy.

CONTACTS AND LOCATIONS:
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
The demographic and biochemical indicators of this study.

REFERENCES:
- [Result] Lauria G, Cornblath DR, Johansson O, McArthur JC, Mellgren SI, Nolano M, Rosenberg N, Sommer C; European Federation of Neurological Societies. EFNS guidelines on the use of skin biopsy in the diagnosis of peripheral neuropathy. Eur J Neurol. 2005 Oct;12(10):747-58. doi: 10.1111/j.1468-1331.2005.01260.x. PMID 16190912
- [Result] Van Acker N, Rage M, Sluydts E, Knaapen MW, De Bie M, Timmers M, Fransen E, Duymelinck C, De Schepper S, Anand P, Meert T, Plaghki L, Cras P. Automated PGP9.5 immunofluorescence staining: a valuable tool in the assessment of small fiber neuropathy? BMC Res Notes. 2016 May 23;9:280. doi: 10.1186/s13104-016-2085-4. PMID 27215701